CLINICAL TRIAL: NCT03441698
Title: Relaxing Effects of Acupuncture, Sham Acupuncture or no Acupuncture, Given by Therapists Delivering Positive or Neutral Communication Regarding Expected Effects
Brief Title: Relaxing Effects of Acupuncture, Sham Acupuncture or no Acupuncture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Västernorrland County Council, Sweden (Other Government)
Collaborators: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Ylva Widgren, Study coordinator, Linkoeping University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Relaxation001
Record Dates: First submitted 2018-02-08; First posted 2018-02-22 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — RE1-silencing transcription factor

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Genuine acupuncture (A) (Experimental): Genuine acupuncture (A) with neutral communication (A1) or positive communication (A2)
  Interventions: Device: Genuine acupuncture (A)
- Sham Acupuncture (B) (Placebo Comparator): Sham acupuncture (B) with neutral communication (B1) or positive communication (B2)
  Interventions: Device: Sham acupuncture (B)
- Rest (C) (Active Comparator): Rest (C) with neutral communication (C1) or positive communication (C2)
  Interventions: Other: Rest

INTERVENTIONS:
Device: Genuine acupuncture (A) — A) Acupuncture is administered bilaterally to the acupuncture point PC6 located two body-inches proximal of the wrist crease, between the tendons of palmaris longus and flexor carpii radialis. Sharp acupuncture needles were inserted into a depth of a half body-inch. The needles are manipulated three times (at the start, middle and end of the treatment session) by twirling and lifting until deqi occurs. Within the groups A, B and C, the participants are randomized to two communication types: 1) neutral communication or 2) strengthened positive communication regarding expected relaxing effects of their treatment, using a standardized communication model.
  Arms: Genuine acupuncture (A)
Device: Sham acupuncture (B) — B) Sham acupuncture is administered bilaterally to a non-acupuncture point two body-inches proximal and one body-inch radial from PC6. The telescopic Park Sham Device was used. The needle looks identical to a real needle, but is blunt and glides upward into its handle instead of penetrating. The marking tubes holds the needle in place. The therapist give an illusion of manipulating the needle by turning it three times until it touched the skin, but no deqi occurs. Within the groups A, B and C, the participants are randomized to two communication types: 1) neutral communication or 2) strengthened positive communication regarding expected relaxing effects of their treatment, using a standardized communication model.
  Arms: Sham Acupuncture (B)
Other: Rest — C) Rest means resting for 30 minutes, either sitting or lying down. Within the groups A, B and C, the participants are randomized to two communication types: 1) neutral communication or 2) strengthened positive communication regarding expected relaxing effects of their treatment, using a standardized communication model.
  Arms: Rest (C)

SUMMARY:
Background: The communication between a patient and clinician may have significant effects on treatment outcomes and one likely mediator of the communication-related treatment effects is patient expectations, as demonstrated by placebo studies in various clinical domains. To investigate the link between patient-clinician interactions and patient expectancy in a clinical setting, acupuncture is suggested an effective method, as acupuncture is a procedure with known non-specific treatment components. As a scene for investigating the importance of expectations on treatment outcomes, the investigators used acupuncture for relaxation effects. It is commonly reported that participants experience a sense of relaxation during acupuncture treatment, yet, it is not known if the effects are related to the specific effects of needling or non-specific effects associated with the treatment procedure.

Aim: To investigate if communication type (positive or neutral) about the expected treatment outcome affected i) participants' expectations, ii) short-term relaxation effects in response to genuine or sham acupuncture or to rest, and to investigate if treatment expectations were related to outcome.

Procedure: Volunteers, i.e. Swedish individuals in general, not part of any specific patient group, are given written and oral study information and are screened for study criteria. The volunteers giving informed consent are randomized to one treatment session a´30 minutes with a) genuine acupuncture or b) sham acupuncture (telescopic non-penetrating needles).

They are compared to a non-randomized reference group that receive no acupuncture, just 30 minutes of rest.

Within the three groups, participants are randomized to 1) positive communication or 2) neutral communication from therapists, regarding expected treatment effects.

Outcome measures: Visual analogue scales (VAS) (0-100 millimeter) measured treatment expectations and relaxation, at baseline two hours before the treatment session, pre treatment (directly before the treatment session) and post treatment (directly after the treatment session). Heart rate, blood pressure, and salivary cortisol are measured pre and post treatment. Primary endpoint is change in relaxation pre to post treatment.

DETAILED DESCRIPTION:
Background: The communication between a patient and clinician may have significant effects on treatment outcomes and one likely mediator of the communication-related treatment effects is patient expectations, as demonstrated by placebo studies in various clinical domains. To investigate the link between patient-clinician interactions and patient expectancy in a clinical setting, acupuncture is suggested an effective method, as acupuncture is a procedure with known non-specific treatment components. As a scene for investigating the importance of expectations on treatment outcomes, the investigators used acupuncture for relaxation effects. It is commonly reported that participants experience a sense of relaxation during acupuncture treatment, yet, it is not known if the effects are related to the specific effects of needling or non-specific effects associated with the treatment procedure.

Aim: To investigate if communication type (positive or neutral) about the expected treatment outcome affected i) participants' expectations, ii) short-term relaxation effects in response to genuine or sham acupuncture or to rest, and to investigate if treatment expectations were related to outcome.

Procedure: Volunteers, i.e. Swedish individuals in general, not part of any specific patient group, are given written and oral study information and are screened for study criteria. The volunteers giving informed consent are blinded randomized, by use of a computerized random table, to one treatment session a´30 minutes with a) genuine manual acupuncture delivered to the traditional acupuncture point PC6 or b) sham acupuncture delivered to a sham acupuncture point at the double distance to the wrist compared to the PC6, using telescopic non-penetrating needles. The acupuncture treatments (genuine or sham) was given by one of nine physiotherapists.

They are compared to a non-randomized reference group that receive no acupuncture, just a treatment of 30 minutes of rest, given by one of three physiotherapists according to a standardized treatment protocol.

Within the three groups (genuine acupuncture, sham acupuncture or no acupuncture, just rest), the participants are randomized to 1) positive communication or 2) neutral communication from therapists according to a standardized treatment protocol, regarding expected treatment effects.

The participants are blinded to type of acupuncture and communication type. The investigator entering data is blinded to treatment type and communication type. The evaluator is blinded to treatment type and communication type.

Outcome measures: Visual analogue scales (VAS) (0-100 millimeter) measure treatment expectations and level of relaxation, muscle tensions and stress at baseline two hours before the treatment session, pre treatment (directly before the treatment session) and post treatment (directly after the treatment session). Heart rate, blood pressure, and salivary cortisol are measured pre and post treatment. Primary endpoint is change in level of relaxation pre to post treatment.

ELIGIBILITY:
Inclusion Criteria:

* minimum age 18 years,
* physical, mental and linguistic capacity to give informed consent, e.g. understand Swedish

Exclusion Criteria:

* previous education in acupuncture therapy, in terms of being an acupuncture therapist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 363 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Change in relaxation from pre to post treatment. | Directly before treatment and directly after treatment.
  Visual Analogue Scale (VAS) 0-100 mm, where 0 is "not relaxed at all" and 100 is "completely relaxed".

SECONDARY OUTCOMES:
Change in treatment expectations | Two hours before treatment, directly before and directly after treatment
  Visual Analogue Scale (VAS) 0-100 mm, where 0 represents "expects treatment to have no effect" and 100 represents "expects treatment to have full effect".
The participant´s Health status | Two hours before treatment
  Euro Qol barometer, 0-100 mm, where 0 represents "worst Health imaginable" and 100 "best Health imaginable"
Change in Heart rate in beats per minute | Directly before treatment and directly after treatment
  Digital wrist blood pressure monitor
Change in systolic Blood pressure in mm Hg | Directly before treatment and directly after treatment
  Digital wrist blood pressure monitor
Change in diastolic Blood pressure in mm Hg | Directly before treatment and directly after treatment
  Digital wrist blood pressure monitor

CONTACTS AND LOCATIONS:
Overall Officials: Anna E Enblom, PhD, Principal Investigator — County council of Östergötland

IPD SHARING:
Plan to Share IPD: No